CLINICAL TRIAL: NCT07285967
Title: A First-in-Human, Randomized, Double-Blinded, Placebo Controlled, SAD and MAD Study in Healthy Participants to Evaluate the Safety, Tolerability, and Pharmacokinetics of YR011 Following Oral Administration.
Brief Title: A First-in-Human SAD and MAD Study in Healthy Participants to Evaluate Oral YR011 Tablet
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Yirui Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: YR011-B01
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Safety; Tolerability; Pharmacokinetics
Keywords: KV1.3; YIRUI pharma; yirui; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- YR011 (Active Comparator): Active arm: Participants receive the investigational drug YR011 at a specific dose.
  Interventions: Drug: Kv1.3 potassium channel blocker (PA032, investigational oral small-molecule drug)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kv1.3 potassium channel blocker (PA032, investigational oral small-molecule drug) — Highly selective Kv1.3 potassium channel blocker (active ingredient: PA032) - oral tablet formulation, administered as single ascending doses or multiple ascending doses (twice daily for 7 days + 1 extra dose on Day 8) under fasting conditions.
  Arms: YR011
Drug: Placebo — The placebo intervention in this study is a matched oral tablet formulationcontaining inactive ingredients (e.g., excipients like microcrystalline cellulose, lactose) with no pharmacological activity.
  Arms: Placebo

SUMMARY:
This is a Phase I clinical trial (protocol number: YR-011-B01) sponsored by Hangzhou Yirui Pharmaceutical Technology Co., Ltd., focusing on the novel oral small-molecule drug YR011 (active ingredient: PA032, a Kv1.3 channel blocker). The trial aims to evaluate the safety, tolerability, and pharmacokinetics (PK) of YR011 in healthy adult participants.

The trial has two stages: Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD), with about 64 participants total (32 per stage). Participants are divided into 4 cohorts per stage (8 people per cohort), randomized 6:2 to receive YR011 or placebo in a double-blind manner. For the SAD stage, 4 dose levels are tested as a single oral dose under fasting conditions; for the MAD stage, 4 dose levels are given twice daily for 7 days plus one extra dose on Day 8.

Key procedures include screening (up to 28 days before enrollment), baseline assessments, drug administration, and follow-up (7 days for SAD, 14 days for MAD). Safety is the primary endpoint (measured by treatment-related adverse events), with secondary endpoints including PK parameters (e.g., plasma concentration, half-life) and dose accumulation. Eligible participants are 18-60 years old, healthy, and able to comply with trial procedures; those with major diseases, drug allergies, or recent medication use are excluded.

The trial follows ICH-GCP and FDA regulations, with a Safety Review Committee overseeing dose escalation and safety monitoring. All data is collected via electronic case report forms (eCRFs) and kept confidential.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase Ⅰ study. The purpose is to investigate the safety, tolerability, pharmacokinetics (PK) of YR011 in adult healthy participants following oral single and multiple ascending dose administration and the recommended dose to be used in the phase Ⅱ study.

This study consists of 2 stages:

Stage 1 (SAD):

The plan is to enroll approximately 32 eligible healthy participants in 4 cohorts. At least 4 cohorts will be studied, with approximately 8 participants in each cohort. Participants will be randomized at a 6:2 ratio to receive YR011 or placebo in a double-blind fashion, i.e. for 8 participants in a cohort, 6 participants will be randomized to receive active drug and 2 participants randomized to receive placebo. Sentinel dosing (1 participant to receive YR011 and 1 participant to receive placebo) will be used in each cohort to ensure adequate safety and tolerability evaluation before administering YR011 or placebo to the remainder of the participants within the cohort. After blinded review by the Safety Review Committee (SRC) of 24-hour post-dose safety and tolerability data from the sentinel group, the remaining 6 participants of each cohort may be dosed, provided that the adverse event (AE) profile in the sentinel participants is considered acceptable.

Four dose levels are planned. However, an additional cohort with a designated dose may be further studied if safety is confirmed in the previous cohorts, as decided by the SRC. The next dose level can only be studied after the SRC reviews the safety data of the previous dose level. For each participant, the drug will be administered once under fasting condition.

Pharmacokinetic blood samples will be collected up to 48 hours after dosing. Participants will be admitted to the Clinical Unit on Day -1, remain at the Clinical Unit until 48 hours post-dose on Day 3 (3 overnight stays), and will return 7 days after dosing for a Follow-up Visit.

The adjustment of the ascending dose will be based on the following rules:

Dose escalation will start from the lowest dose and proceed in the planned escalating sequence. After all participants have received the previous dose of the drug, the investigator and the sponsor will decide whether to escalate to the next dose level. In each dose group of participants, if 1/2 or more participants experience grade 2 or above adverse events (AEs, regardless of the AEs' relation to the study drug), or 1/3 or more participants experience grade 3 or above AEs (regardless of the AEs' relation to the study drug), or one or more participants experience serious adverse events (SAEs, regardless of the AEs' relation to the study drug), dose escalation will be terminated.

After the Stage 1 (SAD) is completed, the sponsor will decide whether to proceed with Stage 2 (MAD), suspend the study for an interim analysis, or terminate the study.

Stage 2(MAD):

There will be approximately 32 eligible healthy participants enrolled in 4 cohorts. Each cohort will include 8 participants. Participants will be randomized at a 6:2 ratio to receive YR011 or placebo in a double-blind fashion, i.e., for 8 participants in a cohort, 6 participants will be randomized to receive active drug and 2 participants randomized to receive placebo. Unlike the single-dose regimen, sentinel dosing within cohorts is not required in the multiple-dose regimen.

Four dose levels as decided by SRC are planned, and will be orally administered twice daily for 7 days, and 1 more dose on the 8th day, followed by a 7-day post-dose follow-up period under fasting condition. However, the dosage and administration method may be modified based on the findings in stage 1 and any new findings in stage 2. Pharmacokinetic blood samples will be collected up to 48 hours after dosing. Participants will be admitted to the Clinical Unit on Day -1, remain at the Clinical Unit until D10 (10 overnight stays), and will return 7 days after dosing for a Follow-up Visit.

The adjustment of the ascending dose will be based on the following rules:

Dose escalation will start from the lowest dose and proceed in the planned escalating sequence. After all participants have received the previous dose of the drug, the investigator and the sponsor will decide whether to escalate to the next dose level. In each dose group of participants, if 1/2 or more participants experience grade 2 or above adverse events (AEs, regardless of the AEs' relation to the study drug), or 1/3 or more participants experience grade 3 or above AEs (regardless of the AEs' relation to the study drug), or one or more participants experience serious adverse events (SAEs, regardless of the AEs' relation to the study drug), dose escalation will be terminated. Safety Review Committee (SRC) The SRC will be comprised of Independent, subject-matter-expert individuals (as qualified by education, training and experience to perform their respective task), not directly involved in the study conduct, for an unbiased review of the trial's emerging safety data and to help inform dose escalation decisions.

A pharmacokinetics expert and other participant matter experts may participate as needed. The SRC will be responsible for ongoing review of safety, tolerability, and clinical laboratory results, and available PK data, and deciding:

1) To escalate to the next planned cohort or alternative dose levels (e.g., lower, intermediate, or higher) in single-dose cohorts (based on a review of available data, including at least 48 hours post-dose safety data and clinical laboratory results from each of the participants in the current cohort); 2) To escalate to the next planned cohort or alternative dose levels (e.g., lower, intermediate, or higher) in multiple-dose cohorts (based on a review of available data, including at least 48 hours post last dose safety data from each of the participants in the current cohort); 3) To add additional dose cohort(s) in either the single- or multiple-dose studies.

4) To decide whether sentinel participants are needed in MAD cohorts. In addition, if ≥ 2 subjects on drug develop the same or similar AE of moderate intensity or if 1 subject develops a severe or serious AE that is considered possibly or probably related to study drug administration, further dosing will be withheld until the SRC investigates the events. Based on this assessment, the SRC will determine if the study should be terminated or continued and whether modification of planned dose levels and/or implementation of additional safety monitoring is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet all the following criteria could be enrolled in this study:

  1. Written informed consent obtained from the participant in compliance with all local legal requirements.
  2. Male or female participant aged between 18 and 60 years (extremes included).
  3. Body mass index (BMI) between 18-32 kg/m2 (extremes included) and body weight less than 120 kg.
  4. Males must use a condom or remain abstinent during the trial and for 3 months after their last dose of study medication. And a fertile man's female partner must not try to become pregnant during the study.
  5. Female participants of childbearing potential must be established on a highly effective method of contraception (The recommended birth control methods are: Implantable (e.g. Implanon(r)), injectable (e.g. Depo-Provera(r)), insertable (e.g. NuvaRing®), Mirena (r) (LNG-IUS)), Combined oral contraceptives pill or progestin-only pill, Evra patch®, Intrauterine device (e.g. ParaGard(r), copper T) or Female sterilization, Male sterilization. The recommended birth control methods must be taken at least 3 weeks prior to screening (i.e., to ensure the contraceptive method has taken effect).) prior to dosing and until 3 months after their last dose in combination with male partner's use of a condom during the trial and for 3 months after the last dose.
  6. Free from any clinically relevant illness or disease that may adversely affect the safety of the participant, or the integrity of the study as determined by medical history, physical examination, safety laboratory, and other assessments.
  7. Participants must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures. Without other intestinal diseases such as irritable bowel syndrome and acute diarrhea due to any infection.

Exclusion Criteria:

* If the participants meet any of the following criteria, they cannot be enrolled in this clinical trial:

  1. Pregnant or lactating women.
  2. Participants with dysphagia.
  3. Severe infections requiring parenteral antibiotics treatment within 4 weeks prior to screening, e.g. sepsis, or severe pneumonia.
  4. Any clinically relevant conditions e.g. cerebral stroke, myocardial infarction, heart failure, unstable angina, and severe heart rate abnormalities within 6 months before screening.
  5. History or presence (within 6 months) of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
  6. Participant has a supine blood pressure outside the ranges of 90 to 140 mm Hg for systolic and 40 to 90 mm Hg for diastolic, confirmed with repeat per PI discretion, at the Screening Visit or Inpatient Check-in (Day -1).
  7. Presence of any renal impairment or dysfunction (i.e. estimated glomerular filtration rate (eGFR)<90 mL/ min).
  8. Presence of hepatic impairment: Child-Pugh A, B or C and/or transaminase levels that are outside the upper normal limit (i.e., Serum bilirubin ≥1.5× upper limit of normal (ULN), ALT or AST levels > ULN).
  9. diagnosis of diabetes regardless the degree of control at screening visit
  10. Hyperthyroidism or hypothyroidism.
  11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
  12. Any major surgery within 6 months of screening.
  13. Participant has a positive test result of HBV (positive HBsAg), HCV (positive anti-HCV), or human immunodeficiency virus I and II (positive anti-HIV I/II), Treponema Pallidum antibody (positive anti-TP) at screening.
  14. Participants with innate or acquired immune system defects.
  15. Participant has a resting heart rate outside the range of 40 to 100 bpm, confirmed with repeat per PI discretion, at the Screening Visit or Inpatient Check-in (Day -1).
  16. Participant has an abnormal (CS) ECG at Screening or Inpatient Check-in (Day -1). Entry of any participant with an abnormal (NCS) ECG must be approved and documented by signature by the Investigator or a medically qualified sub-investigator.
  17. Participant has a QT interval with Fridericia's correction method (QTcF) >450 ms (males) or>470 ms (females) or PR outside the range of 120 to 220 ms, confirmed with one repeat testing at the Screening Visit or Inpatient Check-in (Day -1) Visit; or history of risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome); or the use of concomitant medications that prolong the QT/QTc interval.
  18. Participant has a history of a major psychiatric illness or currently receiving therapy for a psychiatric condition Participant has previously had a seizure or convulsion (lifetime, with the exception of febrile seizures), including absence seizure.
  19. Taken any concomitant medications (including over-the-counter medications such as aspirin, acetaminophen, ibuprofen, herbal [including traditional Chinese medicinal products] or dietary supplements and cough syrup, as well as medicines requiring a prescription) within 14 days or 5 half-lives (whichever is longer), or St John's Wort within 30 days before the study drug administration. etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment- Emergent adverse events (TEAE) | From date of randomization until the last date of the post-treatment follow-up period, up to 44 days after informed consent.
  safety assessment will be based on the incidence of treatment- Emergent adverse events (TEAE) through out the treatment period and until the post-treatment follow-up period

SECONDARY OUTCOMES:
Plasma concentration of YR011 | During treatment period from the first dose to the last dose (up to Maximum of 10 days)
  blood samples will be taken at various timepoints before and after single and multiple dosing of the study drug
Peak Plasma Concentration of YR011 | During treatment period from the first dose to the last dose (up to Maximum of 10 days)
  blood samples will be taken at various timepoints before and after single and multiple dosing of the study drug to assess the Cmax of YR011
Time to peak plasma concentration of YR011 | During treatment period from the first dose to the last dose (up to Maximum of 10 days)
  blood samples will be taken at various timepoints before and after single and multiple dosing of the study drug to assess the Tmax of YR011
Area under the plasma concentration versus time curve (AUC) of YR011 | During treatment period from the first dose to the last dose (up to Maximum of 10 days)
  blood samples will be taken at various timepoints before and after single and multiple dosing of the study drug to assess the AUC of YR011
Half life of YR011 (T1/2) | During treatment period from the first dose to the last dose (up to Maximum of 10 days)
  blood samples will be taken at various timepoints before and after single and multiple dosing of the study drug to assess the T1/2 of YR011

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azam P, Sankaranarayanan A, Homerick D, Griffey S, Wulff H. Targeting effector memory T cells with the small molecule Kv1.3 blocker PAP-1 suppresses allergic contact dermatitis. J Invest Dermatol. 2007 Jun;127(6):1419-29. doi: 10.1038/sj.jid.5700717. Epub 2007 Feb 1. PMID 17273162